CLINICAL TRIAL: NCT02091232
Title: Renal Transplantation Followed By Infusion of T-Regulatory Cells Made With Belatacept Ex-Vivo
Brief Title: Infusion of T-Regulatory Cells in Kidney Transplant Recipients (The ONE Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); University of Regensburg (Other)
Responsible Party: Principal Investigator, James F. Markmann, MD, PhD, Chief, Division of Transplant Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The ONE Study
Record Dates: First submitted 2014-03-13; First posted 2014-03-19 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Kidney Failure, Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: T Regulatory Cell Infusion — After blood is collected from the donor and recipient, the facility will sort out one particular kind of immune cell called a regulatory T cell which is strongly influenced by tolerance induction to minimize (suppress) responses to the donor cells. In this study, these regulatory T cells are the cells which will be given back to the recipient on Day 7 (+3 days) post-transplant.

SUMMARY:
This research study is for patients who are going to receive a kidney transplant from a living donor. After kidney transplantation, it is necessary for transplant recipients to take "immunosuppressive drugs". These drugs work by preventing the body's immune cells from attacking and "rejecting" the new kidney. Taking these drugs long-term may also cause harm to the transplanted kidney. Therefore, the transplant community is very interested in finding ways to decrease immunosuppressive drug treatment and further reduce the risk of kidney rejection. One method to do so is known as "induction of tolerance", which is when the person who receives a transplant has treatment to make their immune cells tolerant to the donor cells.

In this study, we will try to induce tolerance by mixing recipient cells and their donor's cells together with belatacept, an immunosuppressive drug. Belatacept is a protein that attaches to immune system cells, interferes with the immune response and results in tolerance induction.

After we mix the recipient cells with the donor's cells, we will sort out one particular kind of immune cell, called a regulatory T cell, and inject them back into the recipient. Regulatory T cells are the cells that are affected by induction to reduce rejection of donated organs. This method for inducing tolerance has been used in bone marrow transplantation, but this is the first time it is being done in kidney transplantation.

This study is being conducted as part of a unique collaboration of US and EU centers called The ONE Study. The ONE Study centers have agreed to work together using common protocols and procedures but with each testing their own regulatory population for safety and the ability to promote kidney survival. Sharing data among the participating sites will permit a deeper understanding of how and why some treatments might succeed while others work less well.

ELIGIBILITY:
Key Recipient Inclusion Criteria:

* Chronic renal insufficiency necessitating kidney transplantation
* Aged at least 18 years
* Donor is ABO (Blood type) compatible

Key Recipient Exclusion Criteria:

* HIV positive, EBV negative, or suffering from chronic viral hepatitis or tuberculosis
* Previously received any tissue or organ transplant other than planned kidney graft
* Genetically identical to the prospective organ donor at the HLA loci (0-0-0 mismatch)
* Panel Reactive Antibodies (PRA) >20%
* Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non metastatic basal/squamous cell carcinoma of the skin)
* Ongoing treatment with systemic immunosuppressive drugs at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03-02 (Actual); Study Completion 2016-03-02 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility of T Regulatory Cell Infusion in Renal Transplantation | 2 Weeks
  To examine in living donor renal transplant recipients the safety and feasibility of administering T regulatory cells derived from recipient PBMC stimulated with kidney donor PBMC in the presence of costimulatory blockade with belatacept.

SECONDARY OUTCOMES:
T-Reg Measurements | 2 Years
  To measure the presence, potency, and specificity of Treg in the peripheral circulation of kidney transplant recipients.
  This will be done by in-vitro testing of the T-reg cell product and peripheral blood.
Reduction of Immunosuppression | 60 Weeks
  To develop preliminary information on whether administration of the Treg cell product allows a tapering of conventional maintenance immunosuppression within 60 weeks after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jim Markmann, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407
- [Derived] Guinan EC, Cole GA, Wylie WH, Kelner RH, Janec KJ, Yuan H, Oppatt J, Brennan LL, Turka LA, Markmann J. Ex Vivo Costimulatory Blockade to Generate Regulatory T Cells From Patients Awaiting Kidney Transplantation. Am J Transplant. 2016 Jul;16(7):2187-95. doi: 10.1111/ajt.13725. Epub 2016 Mar 11. PMID 26790369
- See also: Related Info — http://www.onestudy.org/